CLINICAL TRIAL: NCT04950101
Title: Prevalence of Anal High-risk Human Papilloma Virus Infection and Abnormal Anal Cytology in Men Who Have Sex With Men Using Pre Exposure Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: HPV Study
Record Dates: First submitted 2021-04-16; First posted 2021-07-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-06

CONDITIONS: Human Papilloma Virus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAS-N (Active Comparator): In this arm the patient without HIV using PrEP will be included
  Interventions: Other: anal sampling
- HAS-P (Active Comparator): In this arm the patient with HIV will be included
  Interventions: Other: anal sampling

INTERVENTIONS:
Other: anal sampling — anal sampling will be performed both in men without HIV and men having HIV in order to see if they have HPV or not

SUMMARY:
The aim of the study is to determine the prevalence of anal high-risk HPV infection and abnormal cytology in HIV uninfected Men who have sex with men (MSM) using PrEP and HIV infected MSM followed-up at the S-kliniek or HRC of the UZ Brussel. 200 participants will be preferably included in the study. The data will be collected using a self-administered questionnaire where socio-demographic characteristics, health-related issues and sexual behavior will be questioned. Also anal canal sampling will be performed for cytological analysis. For the HIV infected MSM, additional information will be extracted from the patient files: CD4+ T-cell count and nadir and duration of combination antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected MSM of 18 years or older using PrEP since at least 3 months
* HIV-infected MSM of 18 years or older

Exclusion Criteria for MSM using PrEP:

* Any intervention in the (peri-) anal region in the past 3 months
* enema within 24h before sampling
* receptive anal sex within 24h before sampling
* current/ongoing peri-anal topical HPV-treatment

Exclusion Criteria for MSM infected with HPV:

* none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of anal high risk HPV infection in MSM using PrEP | 2 year

SECONDARY OUTCOMES:
To compare the prevalence of high risk HPV in MSM using PrEP with that of HIV uninfected MSM not using PrEP | 2 year
  comparation will be done with partially using literature
To compare the prevalence of high risk HPV in MSM using PrEP with that of HIV infected MSM | 2 year
to determine the prevalence of abnormal anal cytology in MSM using PrEP and in HIV infected MSM | 2 year

OTHER OUTCOMES:
to determine the correlation between abnormal cytology and HPV infection in MSM using PrEP | 2 year
To determine possible correlations between the characteristics asked in the questionnaire and the prevalence of high risk HPV infection in both MSM using PrEP and MSM who have HIV | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided